CLINICAL TRIAL: NCT05353062
Title: Bipolar Hemostatic Forceps Versus Standard Therapy by Hemoclip and or Epinephrin Injection as Initial Endoscopic Treatment in Acute Non-variceal Upper GI Bleeding: a Prospective, Randomized Multicenter Study
Brief Title: Bipolar Hemostatic Forceps Versus Standard Therapy in Acute Non-variceal Upper GI Bleeding
Acronym: BeBop
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Theresienkrankenhaus und St. Hedwig-Klinik GmbH (Other)
Collaborators: PENTAX Europe GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BeBop01
Record Dates: First submitted 2022-04-25; First posted 2022-04-29 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Gastrointestinal Hemorrhage
Keywords: Hemostasis, Endoscopic; Randomized Controlled Trial
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Intervention Model Description: Randomized prospective study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard therapy (Active Comparator): Endoscopic therapy with hemoclip +/- injection of epinephrine solution
  Interventions: Procedure: Endoscopic therapy with hemoclip +/- injection of epinephrine solution
- Bipolar hemostatic forceps (Experimental): Endoscopic therapy with bipolar hemostatic forceps
  Interventions: Procedure: Hemostatic therapy

INTERVENTIONS:
Procedure: Hemostatic therapy — Bipolar hemostatic forceps
  Arms: Bipolar hemostatic forceps
Procedure: Endoscopic therapy with hemoclip +/- injection of epinephrine solution — Endoscopic therapy with hemoclip +/- injection of epinephrine solution
  Arms: Standard therapy

SUMMARY:
Bipolar hemostatic forceps will be tested against standard therapy in active, non-variceal, upper gastrointestinal bleeding by a prospective, randomized trial

DETAILED DESCRIPTION:
Patients with active, non-variceal, upper gastrointestinal bleeding usually need an urgent endoscopic treatment. The standard therapy by application of an hemoclip and/or injection of an epinephrine solution is not always successful. Bipolar hemostatic forceps is already being used successfully for the treatment of gastrointestinal bleeding in endoscopic submucosal dissection. Its use in primary endoscopic treatment of non-variceal, upper gastrointestinal bleeding has not been shown yet in a randomized prospective study. Patients with active, non-variceal, upper gastrointestinal bleeding (esophagus or stomach or duodenum) of any cause are randomized (1:1) in standard therapy by combination therapy using an hemoclip and/or injection of an epinephrine solution or experimental therapy by application of the bipolar hemostatic forceps. Cross over-treatment should be tried first in case of failed initial treatment. Rescue treatment by other methods such as application of an Over the Scope Clip (OTSC), angiographic embolization or surgery will be allowed next. All patients receive an additional standard therapy by proton pump inhibitors (PPI). Hypothesis: Endoscopic therapy by application of the bipolar hemostatic forceps is superior to standard therapy regarding technical success and rebleeding rate.

ELIGIBILITY:
Inclusion Criteria:

* Active, nonvariceal, upper gastrointestinal bleeding

Exclusion Criteria:

* Severe coagulopathy unresponsive to blood products transfusions: platelets <20,000; international normalized ratio >3.0; partial thromboplastin time >2 normal

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Successful primary hemostasis | 15 minutes
  Number of participants without further endoscopically visible gastrointestinal bleeding in esophagogastroduodonoscopy
Rebleeding | 30 days
  Number of participants without recurrent endoscopically visible gastrointestinal bleeding in esophagogastroduodonoscopy

SECONDARY OUTCOMES:
Reinterventions | 30 days
  Number of endoscopic reinterventions for gastrointestinal bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Schmitz, MD, Principal Investigator — Helios Kliniken Schwerin
Locations (1):
- Helios Kliniken Schwerin, Schwerin, Germany

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will be available to other researchers on request

REFERENCES:
- [Result] Gralnek IM, Stanley AJ, Morris AJ, Camus M, Lau J, Lanas A, Laursen SB, Radaelli F, Papanikolaou IS, Curdia Goncalves T, Dinis-Ribeiro M, Awadie H, Braun G, de Groot N, Udd M, Sanchez-Yague A, Neeman Z, van Hooft JE. Endoscopic diagnosis and management of nonvariceal upper gastrointestinal hemorrhage (NVUGIH): European Society of Gastrointestinal Endoscopy (ESGE) Guideline - Update 2021. Endoscopy. 2021 Mar;53(3):300-332. doi: 10.1055/a-1369-5274. Epub 2021 Feb 10. PMID 33567467
- [Result] Kataoka M, Kawai T, Hayama Y, Yamamoto K, Nonaka M, Aoki T, Yagi K, Fukuzawa M, Fukuzawa M, Moriyasu F. Comparison of hemostasis using bipolar hemostatic forceps with hemostasis by endoscopic hemoclipping for nonvariceal upper gastrointestinal bleeding in a prospective non-randomized trial. Surg Endosc. 2013 Aug;27(8):3035-8. doi: 10.1007/s00464-013-2860-4. Epub 2013 Mar 7. PMID 23468331
- [Derived] Schmitz D, Thielemann L, Grassmann F. Bipolar haemostatic forceps versus standard therapy by haemoclip + / - epinephrine injection as initial endoscopic treatment in active non-variceal upper GI bleeding: study protocol for a prospective, randomized multicentre trial (BeBop-Trial). Trials. 2023 Jun 15;24(1):407. doi: 10.1186/s13063-023-07394-x. PMID 37322511